CLINICAL TRIAL: NCT03956433
Title: Investigation of the Effect of Daily Consumption of Bioactive Enriched Foods (BEFs) on Biochemical and Anthropometric Markers of the Metabolic Syndrome in Human Volunteers (a Pilot Study)
Brief Title: Effect of Bioactive Enriched Food on Markers of Metabolic Syndrome
Acronym: PATHWAY-27
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Leeds (Other)
Collaborators: The Leeds Teaching Hospitals NHS Trust (Other); AdWare Research Ltd. (Unknown); University of Bologna (Other); European Union (Other)
Responsible Party: Principal Investigator, Samantha Sutulic, Postdoctoral Research Fellow, University of Leeds
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Basic Science
Other Study IDs: PW27_Pilot_Protocol_v1.2
Record Dates: First submitted 2018-01-26; First posted 2019-05-20 (Actual); Last update posted 2019-05-20 (Actual); Status verified 2019-05

CONDITIONS: Metabolic Syndrome
MeSH Terms: conditions — Metabolic Syndrome | interventions — Docosahexaenoic Acids; beta-Glucans; Anthocyanins

STUDY DESIGN:
Intervention Model Description: Five treatment groups, no placebo.
Who Masked: Participant, Investigator
Masking Description: Double-blind
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (5):
- Docosahexaenoic Acid enriched pancakes (Experimental): One portion of pancakes enriched with 250 mg docosahexaenoic acid (DHA) to be consumed daily for 4 weeks.
  Interventions: Dietary Supplement: Ready-made pancakes enriched with docosahexaenoic acid (DHA)
- Beta-glucan enriched pancakes (Experimental): One portion of pancakes enriched with 3 g beta-glucan (BG) to be consumed daily for 4 weeks.
  Interventions: Dietary Supplement: Ready-made pancakes enriched with beta-glucan (BG)
- Anthocyanin enriched pancakes (Experimental): One portion of pancakes enriched with 320 mg anthocyanins (AC) to be consumed daily for 4 weeks.
  Interventions: Dietary Supplement: Ready-made pancakes enriched with anthocyanins (AC)
- DHA+BG enriched pancakes (Experimental): One portion of pancakes enriched with 250 mg docosahexaenoic acid (DHA) plus 3 g beta-glucan (BG) to be consumed daily for 4 weeks.
  Interventions: Dietary Supplement: Ready-made pancakes enriched with docosahexaenoic acid and beta-glucan (DHA+BG)
- DHA+AC enriched pancakes (Experimental): One portion of pancakes enriched with 250 mg docosahexaenoic acid (DHA) plus 320 mg anthocyanins (AC) to be consumed daily for 4 weeks.
  Interventions: Dietary Supplement: Ready-made pancakes enriched with docosahexaenoic acid and anthocyanins (DHA+AC)

INTERVENTIONS:
Dietary Supplement: Ready-made pancakes enriched with docosahexaenoic acid (DHA) — One portion of DHA-enriched pancakes will be eaten each day for 4 weeks.
  Arms: Docosahexaenoic Acid enriched pancakes
Dietary Supplement: Ready-made pancakes enriched with beta-glucan (BG) — One portion of BG-enriched pancakes will be eaten each day for 4 weeks.
  Arms: Beta-glucan enriched pancakes
Dietary Supplement: Ready-made pancakes enriched with anthocyanins (AC) — One portion of AC-enriched pancakes will be eaten each day for 4 weeks.
  Arms: Anthocyanin enriched pancakes
Dietary Supplement: Ready-made pancakes enriched with docosahexaenoic acid and beta-glucan (DHA+BG) — One portion of DHA+BG-enriched pancakes will be eaten each day for 4 weeks.
  Arms: DHA+BG enriched pancakes
Dietary Supplement: Ready-made pancakes enriched with docosahexaenoic acid and anthocyanins (DHA+AC) — One portion of DHA+AC-enriched pancakes will be eaten each day for 4 weeks.
  Arms: DHA+AC enriched pancakes

SUMMARY:
This pilot study will investigate the enrichment type, in pancakes, most effective at improving markers of metabolic syndrome. Ready-made pancakes enriched with either docosahexaenoic acid (DHA), beta-glucan (BG) or anthocyanins (AC), alone or in combination of DHA+BG or DHA+AC, will be consumed for 4 weeks.

DETAILED DESCRIPTION:
There is scientific evidence to support health claims that docosahexaenoic acid (DHA), an omega-3 fatty acid, and beta-glucan (BG), a soluble plant fibre, can help to maintain healthy cholesterol and triglyceride levels. It is also reported that anthocyanins (AC), colour pigments found in many dietary plants, can lower concentrations of low-density lipoprotein (LDL) cholesterol and increase high-density lipoprotein (HDL) cholesterol in dyslipidemic adults. Research studies often focus on bioactives administered as supplements, this study will also investigate the effectiveness of the food matrix. The project addresses the exploitation of bioactive compounds extracted from natural food sources that when added as ingredients to foods and consumed within the common diet, could significantly benefit human health and wellbeing.

ELIGIBILITY:
Inclusion Criteria:

Subjects will be eligible to the pilot study if they present with two to four of the criteria for metabolic syndrome (MetS), at least one of them being alteration of fasting triglycerides or HDL-C cholesterol. MetS is defined when three of the following criteria are met:

* elevated waist circumference (men ≥ 102 cm; women ≥ 88 cm)
* elevated fasting triglycerides (≥ 150 mg/dL)
* reduced fasting HDL-cholesterol (men ≤ 40 mg/dL; women ≤ 50 mg/dL)
* elevated blood pressure (systolic ≥ 130 mmHg and/or diastolic ≥ 85 mmHg) or hypotensive treatment
* elevated fasting glucose (≥ 110 mg/dL)

Exclusion Criteria:

Participants are excluded if three or more clinical criteria for metabolic syndrome are met. Additionally, major exclusion criteria are:

* regular drug therapy with impact on serum lipids;
* diabetes (fasting glucose > 1.26 g/L, or anti-diabetic treatment);
* recent history of cancer or cancer treatment (less than 2 years);
* active or recently diagnosed intestinal malabsorption or disorders associated with malabsorption: Crohn's disease, short bowel syndrome, Pancreatic insufficiency , cystic fibrosis, Tropical Sprue, whipple's disease, chronic pancreatitis, gastrojejunostomy, surgical treatments for obesity, cholestasis, biliary atresia, parasite infections, HIV/AIDS
* familial dyslipidemia;
* use of medication known to cause malabsorption: tetracycline, cholestyramine, thiazide diuretics, aluminum/magnesium hydroxide, colchicine, neomycin, methotrexate, methyldopa, and allopurinol, and laxatives
* illegal drug use, chronic alcoholism or active smoking;
* intensive physical exercise (≥ 5 hour/week);
* consumption of nutritional supplements containing DHA, BG or AC;
* history of allergy or intolerance to any components used in BEFs, celiac disease, lactose intolerance, allergy to milk or egg proteins;
* institutionalised patients, those who lack autonomy to consent or are unable to meet all examinations;
* women who are pregnant, lactating or actively trying to conceive;
* participation in other clinical trials that may impact on outcome;
* subjects deprived of their liberty by judicial or administrative decision.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 35 (Actual)
Dates: Start 2014-09-01 (Actual); Primary Completion 2015-07-04 (Actual); Study Completion 2015-07-04 (Actual)

PRIMARY OUTCOMES:
Fasting triglyceride concentration | Day 1 to Day 28
  Change in fasting triglyceride concentration between baseline and endpoint
Fasting HDL concentration | Day 1 to Day 28
  Change in fasting HDL concentration between baseline and endpoint

SECONDARY OUTCOMES:
Blood pressure | Day 1 to day 28
  Change in systolic and/or diastolic blood pressure between baseline and endpoint
Fasting blood glucose concentration | Day 1 to day 28
  Change in fasting blood glucose concentration between baseline and endpoint
Waist circumference | Day 1 to day 28
  Change in waist circumference between baseline and endpoint
Body mass index | Day 1 to day 28
  Change in body mass index between baseline and endpoint

CONTACTS AND LOCATIONS:
Locations (1):
- University of Leeds, Leeds, West Yorkshire, United Kingdom

IPD SHARING:
Plan to Share IPD: No